CLINICAL TRIAL: NCT03550183
Title: Safety and Efficacy Investigation of Patients With Parkinson's Disease by Transplantation of Umbilical Cord Derived Mesenchymal Stem Cells
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Therapy in Parkinson's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hebei Newtherapy BIo-Pharma technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shengjun An, Principal Scientist & Professor, Hebei Newtherapy BIo-Pharma technology Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18967728D
Record Dates: First submitted 2018-05-11; First posted 2018-06-08 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mesenchymal stem cells (Experimental): Selected patients with Parkinson's disease were randomly divided into a therapy group and a control group. Umbilical Cord Derived Mesenchymal Stem Cells(UC-MSCs) at a dose of 10-20 million by intravenous infusion.Patients in the therapy group treated once a week with UC-MSCs. Each course of treatment Lasted 3 weeks.
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — Patients with PD in the therapy group were given UC-MSCs by intravenous infusion and conventional therapy. There was only conventional treatment in the control group. All patients after treatment for 1 month, 3 months, 6 months and 12 months were evaluated respectively the curative effect.

SUMMARY:
This study is to evaluate the safety and efficacy of Umbilical Cord Derived Mesenchymal Stem Cells transplantation in Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative movement disorder，which mainly shows up in the elderly. And there is as yet no effective drug treatment. Umbilical cord derived mesenchymal stem cells (UC-MSCs) derived from mesoderm owns strong proliferation ability and multiple differentiation potential. The investigators used UC-MSCs via intravenous infusion to treat PD. With different durations of follow-up, the investigators cleared therapeutic effect, the quality of life and prognostic implications of UC-MSCs on PD through the Unified Parkinson's Disease Rating Scale (UPDRS), revised Hoehn-Yahr（H-Y） staging, Mini-Mental State Examination (MMSE), Hamilton depression scales 24 (HAMD 24), Hamilton Anxiety Scale 14 (HAMA 14) and Clinical Global Impression (CGI). In this research, the investigators seek new therapeutic approaches for PD, and provide clinical evidences for the clinical application of UC-MSCs in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 40 to 60 years, and no limitation of gender.
2. Diagnosis of primary Parkinson's disease(PD) according to Movement Disorder Society (MDS)-PD criteria established in 2015.
3. Hoehn-Yahr Stages from I to IV stage.
4. Drugs for anti Parkinson's disease have been taken over 28 days before entering the group.
5. MMSE score≥25
6. No antidepressant or antipsychotic drugs were received within 2 weeks.
7. Understanding and willingness to sign a written informed consent document.

Exclusion Criteria:

Patients with PD have to be disqualified from this study if any of the following is applicable.

1. Patients with psychiatric history, but depression.
2. Suicidal tendency or behavior of patients.
3. Patients with severe cognitive impairment, chronic organ failure or malignant tumor.
4. The value of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) was 1.5 times higher than that of the normal reference; or leucocyte count<1000/μl.
5. Pregnancy and lactating women.
6. The patient is taking part in other drug tests, or received other research medication within 90 days before entering the group.
7. Patients who had quit our study could not enter it again.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2022-10-10 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes of the Unified Parkinson's Disease Rating Scale (UPDRS) | Post cell transplantation: 1, 3, 6, 12months
  The UPDRS was assessed to identify the severity of PD. It includes the four-scale structure with a reorganization of the various subscales. This four-scale structure are (Part I) nonmotor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (18 items), and (Part IV) motor complications (six items). Each subscale now has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe.

SECONDARY OUTCOMES:
Changes of in the Hoehn and Yahr staging | Post cell transplantation: 1, 3, 6, 12months
  Hoehn and Yahr (H-Y) staging was used to determine the stage of PD based on clinical findings and functional disability. In H-Y staging is a rating scale measured in an ordinal level.
Changes of the Mini-Mental State Examination (MMSE) | Post cell transplantation: 1, 3, 6, 12months
  The MMSE was used to measure cognition. This test consists of 2 parts: language and performance. Its total score can range from 0 to 30, with a higher score indicating better function.
Changes of the Hamilton depression scales 24 (HAMD 24) | Post cell transplantation: 1, 3, 6, 12months
  The HAMD 24 is used to assessed the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. There are 24 items in the HAMD 24.
Changes of the Hamilton Anxiety Scale 14 (HAMA-14) | Post cell transplantation: 1, 3, 6, 12months
  The HAMA-14 is used to assessed the anxiety symptoms. Its total score can range from 0 to 56. Lower score represents a better outcome.
Adverse reaction | Post cell transplantation: 1, 3, 6, 12months
  Adverse reaction including temperature changes,the change of blood pressure,allergy and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Xiqing Chai, Doctor, Study Chair — Hebei Chemical & Pharmaceutical College; Ping Gu, Doctor, Study Director — The First Hospital of Hebei Medical University; Hongxu Chen, Master, Study Director — The First Hospital of Hebei Medical University
Locations (1):
- Hebei Newtherapy BIo-Pharma Technology Co., Ltd, Shijiazhuang, Hebei, China